CLINICAL TRIAL: NCT05951439
Title: Effects of Combined Creatine Monohydrate and β-Hydroxy-β-Methylbutyrate Supplementation on Body Composition, Physical Performance, Quality of Life, Oxidative Stress, and Inflammation in Physically Active Older Individuals Who Underwent a Comprehensive Fitness Program: A Randomized Crossover Clinical Trial
Brief Title: Effect of Creatine+HMB Supplementation in Physically Active Older Adults
Acronym: CRESHARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Burgos (Other)
Responsible Party: Principal Investigator, Juan Francisco Mielgo, Assistan Professor, Universidad de Burgos
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: IR 24/2023
Record Dates: First submitted 2023-06-18; First posted 2023-07-19 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2024-12

CONDITIONS: Aging; Sarcopenia; Nutrition, Healthy
Keywords: aging; sarcopenia; nutrition; HMB; creatine; exercise; GAA
MeSH Terms: conditions — Sarcopenia; Motor Activity

STUDY DESIGN:
Intervention Model Description: Cross Randomized double-blind study
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group 1 (Experimental): CRE-HMB mixture
  Interventions: Dietary Supplement: CRE + HMB
- Intervention Group 2 (Placebo Comparator): placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: CRE + HMB — 3 g/day of CRE and 3 g/day of HMB
  Arms: Intervention Group 1
Dietary Supplement: Placebo — 6 g/day of inulin
  Arms: Intervention Group 2

SUMMARY:
Sarcopenia (SAR) is the loss of muscle strength and mass caused by aging. It is accompanied by a progressive decline in physical and cognitive abilities, increasing the risk of falls. This loss of muscle mass leads to pathophysiological changes at the neuromuscular and tendon levels as a consequence, among others, of alterations in the balance between protein synthesis and degradation, inflammation (INF), or alterations in the anabolic/catabolic state (ACS). These alterations are caused by oxidative stress (OS), when reactive oxygen species-toxic metabolites produced by cells using oxygen-exceed the defensive capacity of the antioxidant system.

Therapeutic strategies to modulate SAR are based on exercise and nutrition programs. Multicomponent physical exercise programs have shown improvements in parameters related to sarcopenia. Likewise, the use of nutritional supplements such as creatine (CRE) has demonstrated improvements in muscle function in older adults. CRE may reduce INF and OS in the general population.

On the other hand, beta-hydroxy-beta-methylbutyrate (HMB) also appears to improve muscle function in older adults by promoting myogenesis. However, the effects of these supplements in older adults have only been observed when used in isolation. In this regard, our research team observed that a 10-week regimen combining 3 g/day of CRE + 3 g/day of HMB (CRE-HMB) improved muscle recovery (better ACS) and physical performance in athletes subjected to high muscle wear. However, to date, it has not been determined whether this combination improves muscle function, OS, INF, and ACS in women with SAR.

Therefore, the working hypothesis is that the CRE-HMB combination could improve muscle function and physical performance, as well as OS, INF, and ACS in individuals with high muscle loss, such as those with SAR. Thus, a randomized double-blind crossover study is proposed to analyze the effect of 12 weeks-6 weeks of intervention + 3 weeks of washout + 3 weeks of intervention-of co-supplementation with 3 g/day of CRE + 3 g/day of HMB (CRE-HMB), combined with 4 sessions/week of multicomponent physical exercise, on muscle function, OS, INF, and ACS in 40 physically active men and women over 60 years of age. These 40 participants will be divided into two groups of 20 (20 in the placebo group and 20 in the CRE-HMB group).

At the assessment points (baseline, at 6 weeks, after the 3-week washout period, and after another 6 weeks), body composition, nutritional intake, muscle strength, and performance tests will be evaluated. Blood samples will also be collected to determine biochemical markers of OS, INF, and ACS.

It is expected that CRE-HMB co-supplementation for 6 + 6 weeks, together with multicomponent physical exercise, in physically active older adults will improve muscle strength, muscle mass, and performance. Additionally, improvements in OS, INF, and ACS levels are anticipated.

DETAILED DESCRIPTION:
Study design: Cross-over, controlled, randomised, double-blind study approved by the Bioethics Committee of the University of Burgos (ref. IR 24/2023).

Duration: 15 weeks in total. 6 weeks of intervention, 3 weeks of rest and another 6 weeks of intervention.

Supplementation: 3 g of creatine monohydrate + 3 g of beta-hydroxy-beta-methylbutyrate (HMB).

Control: 6 g of inulin (placebo). Recruitment sessions (T0): 15/8/2024; First meeting with potential participants to explain the study. Reasons, objectives, inclusion and exclusion criteria, study discipline, duration, control dates, resolution of doubts and concerns, etc. They were provided with an information document, a form to collect social data and another with the informed consent form. A first group of 40 people was formed, 15 women and 25 men.

Between September and October 2024, the study's registered dietitian-nutritionist conducted individual nutritional consultations with all participants. Surveys were conducted on food consumption frequency, adherence to the Mediterranean diet, dietary habits, training, sports, pathologies, medications, supplementation, social circumstances, etc. The inclusion and exclusion criteria, the study protocol, randomisation, how to take the supplements, the timing of the tests, how to keep exercise and nutrition records, and the premises of nutrition and exercise (no changes in diet or exercise habits throughout the study) were explained again, as well as who to contact in case of doubt, etc.

Inclusion criteria: all individuals over the age of 60 who performed Comprehensive Physical Conditioning training for a minimum of 120 minutes per week were included. They did not take the study supplement or any other supplement related to performance or muscle development. They did not have heart, liver or kidney disease. Nor did they have musculoskeletal conditions or injuries that required the use of anti-inflammatories during the study. They agreed to the study protocol and signed the informed consent form.

Exclusion criteria: all individuals who were not in the age range studied were excluded. They did not meet the minimum weekly Comprehensive Physical Conditioning training requirement. All those who had suffered from or were being treated for heart, liver or kidney conditions. Those who were being treated with NSAIDs. Those who refused to stop taking supplements and/or follow the study protocol. Ten people were excluded, five women and five men.

Participants: finally, 30 volunteer participants (n=60) were recruited, 10 women (n=20) and 20 men (n=40) over the age of 60 who were doing multi-component training. All signed the informed consent form. They had no impediments to complying with the study protocol.

Randomisation: each participant was randomly assigned to one of the two intervention groups by an independent researcher. Block randomisation was used, ensuring that each group had an equal number of participants and an equal number of men and women. Intervention group (n=15); 3g of CREATINE + 3g of HMB. Control group (n=15); 6g of Inulin.

Timing: the study was divided into 3 stages with 4 controls.

* Stage 1: 6 weeks of intervention. The first control was performed at the beginning on 8/11/2024 (T1) and the second at the end of the 6 weeks on 20/12/2024 (T2).
* Stage 2: 3 weeks of rest or wash-out (T2-T3). 21/12/2024 to 9/1/2025.
* Stage 3: 6 weeks of intervention. The third check-up was performed at the beginning on 10/1/2024 (T3) and the fourth check-up was performed on 21/2/2025 (T4).

Physical exercise during the intervention: the physical conditioning programme implemented in this study was designed in a comprehensive and advanced manner (IPC), with an approach that included both multifunctional and/or multicomponent circuits and specific strength/power interval training sessions (sets). The strategic combination of these modalities is supported by scientific literature as one of the most effective ways to simultaneously improve strength, power, aerobic endurance, and functional capacity in older adults, while respecting the principles of individualisation, progression, variability, transfer, and specificity. This combination allowed for the simultaneous training of several physical abilities, adapting the intensity and exercises to the individual needs of the participants, maximising the benefits in basic physical abilities: strength, endurance (muscular and cardiovascular), speed (movement, execution and reaction), flexibility (static and dynamic), mobility (ROM and RAM) and complex physical abilities: coordination, balance, precision, proprioception, etc.

All participants underwent guided and personalised Integral Physical Conditioning (IPC) training at a frequency 4 weekly sessions lasting 60 minutes with a self-perceived intensity of at least 6 and at most 9 on the modified BORG scale (1-10), combined with activities specific to each subject, non-guided, of low or moderate intensity and oriented towards recreation and/or master competition (swimming, cycling, walking or hiking, paddle tennis, dancing, etc.), carried out on days off from guided training. These activities were practised 1 to 3 times per week, for 20 to 120 minutes per session, and with a self-perceived intensity between 3 and 6 on the modified BORG scale (1-10).

* IPC training:

  * Frequency: 4 sessions per week.
  * Duration: 60 minutes.
  * Equipment: body weight, barbells, dumbbells, kettlebells, elastic bands, medicine balls and giant balls, Bosu balls, plinths, plyometric boxes, pulleys, ballet and calisthenics bars, rings, landmines, sleds, tyres, ropes (climbing and battle), IndoBoards, coordination ladders, Vertimax, stationary bikes, rowing machines, ellipticals, Nautilus-type weight machines, among others.
  * Teaching methodology: direct instruction and assignment of tasks.
  * Type: individualised training.
  * Organisation: Horizontal and Vertical.
* Session structure:

  * Warm-up (5-12 minutes): included mobility, balance, coordination and dynamic flexibility exercises, organised into blocks of progressive difficulty and effort. It was carried out over 10 metres, alternating between walking and jogging. It began with descending joint mobility (optimal ROM) during walking, progressing to more global and demanding exercises (rapid movements, throws, pushes, pulls, turns, push-ups, position changes, jumps, etc.), activating the cardiorespiratory and metabolic systems. It ended with active stretching and a 2-3 minute break for hydration and recovery.
  * Main Part (40-50 minutes): the intensity was medium, medium-high and high. Multifunctional circuits and interval training were implemented, with horizontal and/or vertical organisation, in the same session or in different sessions, depending on the objectives of the microcycle.
* Multifunctional/Multicomponent Circuit Training: Circuit training sessions were structured to work on different physical abilities at the same time. Each station in the circuit was designed and sequenced to address a specific component, such as muscle strength, muscular and cardiovascular endurance, speed (movement, execution and reaction), balance, flexibility, joint mobility and coordination. In this way, participants performed combined exercises that involved both strength work with weights, elastic bands, medicine balls, body weight, equipment, etc., as well as speed, endurance, flexibility and mobility, balance and coordination exercises. This approach allows for medium-high/high intensity work throughout the circuit, maintaining cardiovascular demand while optimising different abilities at each station. This type of training not only optimises training time but also increases cardiovascular demand, improving metabolic efficiency and aerobic endurance. In addition, the variability in the exercises fulfils a fundamental principle of training and prevents monotony, favouring adaptation to several different stimuli simultaneously, resulting in better functionality and physical condition.
* High-Intensity Interval Training: High-intensity interval training (HIIT) sessions adapted to the participants' abilities were incorporated. This method involves alternating periods of intense effort with periods of rest or low-intensity activity. It also involves horizontal and vertical organisation. Interval training is highly effective in improving both aerobic and anaerobic capacity and has been shown to be particularly beneficial in increasing endurance capacity, body composition (MLG) and improving cardiovascular function, even in older adult populations. In this protocol, the high-intensity phases were adjusted according to the individual needs of the participants, ensuring that the efforts were challenging but safe.
* Strength Training: in addition to functional circuits, specific strength training sessions were included with horizontal and vertical organisation. Progressive overload (weights, machines, bands, body weight, etc.) was used to strengthen the main muscle groups, focusing on developing maximum muscle strength and localised muscle endurance. Participants performed sets of exercises focused on developing strength in large and small muscle groups, following a priority criterion based on muscle size, from largest to smallest. Work was done by zones, hemispheres and/or specific muscles. This modality allowed for greater concentration on improving maximum strength, using progressive weights and more structured sets, which complemented the benefits of circuit training and promoted muscle adaptation. This type of training is essential for preventing sarcopenia, improving body composition (LBM and BMR) and strength, thereby helping to maintain muscle health and functional independence.
* Power training: sessions were conducted with high-speed exercises (medicine ball throws, explosive lifts, adapted ballistic movements, plyometric jumps, etc.) with the aim of improving explosive strength and reaction speed. These movements, performed at high speed, were adapted to the participants' abilities, ensuring that the efforts were safe but challenging. Power training has direct benefits on improving explosive strength and reaction speed, which is essential for fall prevention and maintaining functional independence. In addition, incorporating this type of training promoted an improvement in neuromuscular efficiency, optimising the participants' ability to generate force quickly in everyday situations. This combined methodology optimises the development of functional strength and mobility and improves the participants' reaction capacity and agility.
* Cardiovascular endurance training: specific blocks of aerobic work (brisk walking, stairs, cycling, adapted running or elliptical training) were incorporated, both continuously and intermittently. This improved VO₂ max, cardiometabolic health, and exercise tolerance, which are critical aspects of maintaining the overall health of older adults. Circuit training was also combined with other skills. In addition, participants practised moderate-intensity outdoor aerobic activities on their own (walking, hiking, swimming, cycling, paddle tennis, golf, dancing), 1 to 3 times a week, for 20 to 120 minutes, at self-perceived intensities of 3 to 6 (modified Borg).
* Joint mobility (ROM/RAM): specific active and dynamic mobility exercises were incorporated, both as part of the warm-up and within the circuits. Full range of motion in the hips, spine, shoulders, ankles and other key joints was stimulated through functional exercises and dynamic stretching. This component is essential for maintaining functional flexibility, improving movement efficiency and reducing joint stiffness, promoting autonomy in everyday activities.
* Training loads: the quantitative and qualitative factors of the training varied according to the objectives of the microcycle and the type of training. The training heart rate (THR) was calculated using the Karvonen formula, 1RM estimated using Brzycki formula.
* Multicomponent Circuits and HIIT: intensity from 40% to 100% of Training Heart Rate (THR)= 4-10 RPE. Rest periods of 10 to 30 seconds between exercises, and 0 to 2 minutes between rounds. Three to ten rounds were performed, with 5 to 100 repetitions or time-based work (10 seconds to 5 minutes).
* Strength training: intensity of 60% to 90% of estimated 1RM = 6-9 RPE, 3 to 6 sets of 6 to 12 repetitions. Rest periods of 1 to 3 minutes depending on the objective. The analytical work was organised as follows
* Power training: intensity of 20% to 80% of estimated 1RM = 2-8 RPE, 3 to 9 sets of 1 to 5 repetitions. Rest periods of 30 seconds to 3 minutes depending on the objective. Global movements and weightlifting exercises were used: Snatch and clean and jerk.
* Endurance training: intensity of 40% to 60% THR = 4-6 RPE., 1 to 4 sets of 3 to 20 minutes. Breaks of 0 seconds to 1 minute, depending on the method used (continuous or interval) and the objectives.

  * Cool down (5-15 minutes): simple, short games (3-5 minutes), stretching using different methods depending on the session objectives (proprioceptive neuromuscular facilitation, dynamic and/or static stretching, myofascial self-massage with a roller, etc.), breathing and relaxation exercises.

Nutrition and supplementation during the intervention: all participants were instructed to maintain their eating habits without making any changes to their usual diet throughout the intervention. In addition, they were asked to discontinue any previous supplementation to avoid interference with the study protocol. Assessments of food consumption frequency, adherence to the Mediterranean diet, and dietary habits were carried out to verify that there were no changes in diets or habits during the study, as well as to explain the possible relationship between these and the parameters studied.

Supplement delivery: The study supplementation was administered mixed with yoghurt or fruit juice, half an hour before bedtime. The supplement was delivered at the end of the T1 and T3 checks. Each participant received a box containing 42 individual bags with 6 grams of product: either 3 g of creatine + 3 g of HMB or 6 g of placebo (inulin). The allocation was blinded to both the participants and the team member responsible for delivery. Along with the supplement, an information sheet and a control form were included to record the training loads performed during the intervention. These forms were collected and reviewed at the T2 and T4 check-ups.

Data collection and measurement: Data collection and processing were managed through the creation and distribution of Data Collection Notebooks (DCNs) among the research team members. To ensure data quality and traceability, a Data Management Plan and a Statistical Analysis Plan were designed to guide all phases of the process. A specific electronic database was created to enter the follow-up information for each participant, with integrated verification tools to minimise errors during data entry. The physical DCRs were stored and safeguarded by the research team and used as the official source for the preparation of the final report. All information was accurately recorded following the guidelines of the research protocol and the DCR. The data was then transferred to the digital database on a computer dedicated exclusively to the study, protected by IT security systems.

Confidentiality and regulatory compliance: Current data protection legislation was fully complied with, including Organic Law 3/2018 of 5 December on the Protection of Personal Data and Guarantee of Digital Rights, as well as Regulation (EU) 2016/679 of the European Parliament and of the Council of 27 April 2016 (GDPR). Each participant was identified by a unique alphanumeric code, without including any data that would allow their direct identification. The correspondence between the code and the personal data was stored in a separate file, protected by a password and computer security systems. Only authorised personnel had access to this information, thus ensuring the confidentiality and anonymity of the data throughout the study.

General tests and functional assessments

* Blood sampling: performed in the antecubital vein by the research team's laboratory technician. At least three hours after the last meal and 24 hours without physical exercise (previously informed). Ten millilitres were extracted into two tubes using the Vacutainer™ system (BD, Franklin Lakes, NJ) with EDTA as an anticoagulant, which were centrifuged on the same day of collection at 3000 rpm for 10 minutes at 4 °C to obtain a 5 ml tube of plasma, which was frozen at -80°C for storage until subsequent shipment and analysis at the University of Burgos (UBU) laboratory.
* Body composition: participants were assessed using the Tanita MC-580 electrical bioimpedance analysis (BIA) body analyser and Suitbiological 8.0 software. Measurements were also taken of the circumference of the contracted arm, waist, hips and thigh .

The MC-580 measured segmental body composition using multiple frequencies (5, 50, 250 kHz) and provided: Body weight, Body Mass Index (BMI), Total fat mass (%) and in kg, Visceral fat, Total and segmental muscle mass (arms, legs, trunk), Estimated bone mass, Total body water, Basal metabolic rate (BMR), Sarcopenia index, Estimated metabolic age, Health indices (Tanita's proprietary 'Body Quality Index') and Left-right balance in muscle mass. The conditions were controlled according to the manufacturer's criteria because the accuracy of these devices can be affected by factors such as hydration, recent food intake, previous exercise and the menstrual cycle, so it was essential to take measurements under controlled conditions. In addition, the reliability of this model has shown consistent results in validation studies, especially when standardised measurement protocols are followed. Several studies have demonstrated high reproducibility in body composition measurements, with intraclass correlation coefficients (ICC) greater than 0.90 for variables such as fat mass and fat-free mass. Comparisons with reference methods such as DEXA have shown moderate to high correlations (r = 0.80 to 0.95), although with a tendency to slightly underestimate body fat percentage in certain population groups (obese).

ALM_BMI, an index calculated by dividing appendicular lean mass (ALM) by body mass index (BMI), was calculated manually. It is used to assess relative muscle mass adjusted for body size and has been proposed as a useful clinical indicator for the diagnosis of sarcopenia and for predicting functional and metabolic risks in older adults. BSA, or body surface area, was also calculated, which is an estimate of the total area of the external surface of the human body. It is expressed in square metres (m²) and is commonly used in clinical settings to adjust drug doses (especially in oncology), assess physiological functions (such as glomerular filtration or cardiac output), and compare physiological variables between people of different body sizes.

* Vital signs and physiological parameters: all participants had their blood pressure (BP), systolic (SBP) and diastolic (DBP) pressure, and pulse measured using an OMROM model M6-A6 digital oscillometric sphygmomanometer. Three measurements were taken in a seated position, with the arm flexed and supported, and the sphygmomanometer placed at heart level. The best measurement was recorded. Oxygen saturation (%O2) was measured using a BRAUN YK-81CEU clip pulse oximeter. The maximum expiratory force (MEF) was measured using a Pinnacle Peak Flow mechanical expiratory flow meter. Three attempts were made, and the best measurement was recorded.
* Assessment of strength and physical condition:
* Grip strength: measured with a validated JamarÒ plus hydraulic hand dynamometer. Grip strength (kg) was measured in a seated position, with the elbow bent at 90° and the wrist in a neutral position. Participants were asked to apply maximum grip strength in three attempts (30 seconds rest) with their dominant hand, taking the highest value.
* Isometric strength of legs and back: a BASELINE traction dynamometer (back and leg dynamometer) with adjustable handle and base platform was used. The objective was to assess the maximum isometric strength of the back and leg extensor muscles (kg). The subject stood with their feet shoulder-width apart on the dynamometer platform. The legs were slightly bent and the back was in a neutral, inclined position. The dynamometer was adjusted so that the subject could grasp the handle with their arms fully extended downwards (near the knees). The subject was asked to pull the handle upwards, using their back and leg strength, without bending their arms or leaning their trunk backwards. The movement was isometric; force was applied without visible displacement. The contraction lasted about 3 to 5 seconds. Two attempts were made with at least 30 seconds of rest between them. The maximum value achieved was recorded. High test-retest reliability (intraclass correlation coefficients, ICC > 0.94-0.98).
* Isometric arm flexion strength: a BASELINE traction dynamometer with adjustable handle and base platform was used. The objective was to assess the maximum isometric strength of the upper body (kg), specifically the arm flexor muscles (biceps). The subject stood with their feet shoulder-width apart on the dynamometer platform. Their legs were slightly bent and their back was straight and upright. The dynamometer was adjusted so that the subject could grasp the handle with their arms bent at 90°, elbows close to the body and wrists in a supine position. The subject was asked to pull the handle upwards, exerting force with their arms, without leaning the trunk backwards or using momentum. The movement was isometric; force was applied without visible displacement. The contraction lasted about 3 to 5 seconds. Two attempts were made with a 30-second rest between them. The maximum value achieved was recorded. The test-retest reliability of the isometric biceps strength test with a dynamometer is high, with intraclass correlation coefficients (ICC > 0.90) reported in different studies.
* Short Physical Performance Battery (SPPB): Three tests were performed: balance, walking speed (4 m) and chair rise (5 repetitions x time) to assess physical functioning. Each test was scored from 0 to 4 (0 - cannot be completed and 4 - highest level of performance). Total scores range from 0 to 12 (highest level of physical performance). The times and scores for each test were recorded separately and the total score was recorded.
* Timed-up-and-go (TUG): used to assess mobility, balance and agility. The time taken to stand up from a chair, walk 3 metres, turn around, return and sit down was recorded.
* Seated dumbbell arm curl test: the dynamic strength of the arm flexor muscles was measured.

The participant sat on a chair without armrests, with their back straight and their feet flat on the floor. They held a dumbbell in their dominant hand with their palm facing upwards and their arm fully extended down at their side. In 30 seconds, the participant completely flexed their elbow, bringing the dumbbell towards their chest without moving their shoulder, and then extended it again.

Complete repetitions were counted. A 2 kg dumbbell was used for women and a 4 kg dumbbell for men. High test-retest reliability (CCI > 0.80-0.90) in different studies with older adults.

* 30-second push-up test: this was performed to assess the muscle strength and endurance (push) of the upper body (mainly pectorals, deltoids and triceps) and the stabilising strength of the lumbar-abdominal girdle. It consisted of performing as many push-ups as possible in 30 seconds from a plank position. The participant is placed in a high plank position with arms extended, hands shoulder-width apart, and body aligned from ankles to head. Each push-up must be performed with a full range of motion: lower the chest close to the floor (about 5-8 cm) and fully extend the elbows when rising. Only correctly executed repetitions were counted and recorded. High test-retest reliability (ICC > 0.85) in physically active older populations.
* 30-second supine trunk flexion test (Crunch Test): the objective was to assess abdominal muscle endurance. The subject lay supine with knees bent at 90° and feet flat on the floor and arms crossed over the chest. At the evaluator's signal, the subject performed as many trunk flexions as possible in 30 seconds. A repetition was counted as valid when the shoulders clearly lifted off the floor without lifting the lower back and returned to the starting position. The total number of correct repetitions was recorded. High test-retest reliability (CCI > 0.85).
* Isometric pull-up strength test (Flexed Arm Hang Test): used to assess the isometric strength and muscular endurance of the upper body, especially the arms, shoulders and back. Hanging from the bar, keep your head above the bar for as long as possible. The subject stands under a fixed horizontal bar, such as a pull-up bar. With the help of a bench or assistance, they position themselves with their elbows bent and their chin above the level of the bar. The palms may be pronated. The stopwatch starts when the person is suspended without assistance, with their feet completely off the ground. The test ends when the chin falls below the bar, the arms are extended, or the subject lets go. High test-retest reliability (ICC > 0.85) .
* 400-metre walk test: assessed mobility, endurance and maximum oxygen consumption (VO2). A line of cones is placed 20 metres apart, around which participants must walk 10 times as fast as possible. They may stop, but not sit down. Only one attempt is allowed. The total time elapsed is recorded. High test-retest reliability (CCI > 0.90).

Quality of Life Assessment: The WHOQOL-BREF test was used in all controls (T1, T2, T3 and T4). This questionnaire is a shortened version of the WHOQOL-100 questionnaire, developed by the World Health Organisation (WHO) to assess quality of life. It is one of the most widely used instruments internationally due to its psychometric robustness, cross-cultural applicability and brevity. High test-retest reliability (ICC > 0.69-0.91).

Nutritional assessment: the nutritional analysis of the participants was performed using a multidimensional approach that included both food consumption frequency (T1 and T4) and adherence to the Mediterranean diet (T1, T2, T3, T4) and dietary habits (T1 and T4). The participants' dietary data were obtained through surveys and interviews, which provided information on the frequency and quantity of key food consumption. The content of macronutrients (carbohydrates, proteins and fats) and micronutrients (vitamins and minerals) was analysed, as well as the consumption patterns of foods rich in antioxidants, healthy fats and fibre.

- Food Frequency Questionnaire (FFQ): Participants' dietary habits were assessed using a Food Frequency Questionnaire (FFQ) specifically developed for physically active older adults, which took into account consumption over the previous 3 months. This instrument included 24 food items organised into functional groups (dairy, meat, fish, cereals, fruit, vegetables, healthy fats, beverages and processed foods) and was validated by experts in nutrition and exercise science. High test-retest reliability (CCI > 0.85).

Consumption frequency was recorded according to standardised categories: never or almost never, 1-3 times/month, 1 time/week, 2-4 times/week, 5-6 times/week, once/day and 2 or more times/day, which were assigned quantitative values for weekly frequency (e.g., 'once/day' = 7 times/week), according to methodological protocols previously reported in the literature.

Nutritional analysis was performed using an automated template in Microsoft Excel, which allowed for:

* Automatic coding of the recorded frequencies.
* Estimation of weekly intake of key nutrients, including protein, fibre, vitamin C, omega-3 fatty acids, antioxidants, healthy fats, creatine, β-hydroxy-β-methylbutyrate (HMB), sodium, sugars and vitamin D.
* Obtaining a total summary of nutrients per participant and per group. Nutritional composition estimates per serving were obtained from national food composition databases, the Spanish Food Composition Database (BEDCA). This approach allowed us to establish relationships between the subjects' dietary patterns and the main outcomes of the study, in line with the proposed objectives.
* Mediterranean Diet Adherence Survey (PREDIMED): to assess adherence to the Mediterranean diet, the validated questionnaire from the PREDIMED study was used. High test-retest reliability (CCI > 0.70). This questionnaire consists of 14 items that explore the frequency of consumption of foods characteristic of the Mediterranean diet, such as olive oil, fruit, vegetables, fish, nuts, and the consumption of red meat and sugary drinks. Responses are classified into two categories: 'YES' (indicating adherence) and 'NO' (indicating non-adherence), with values assigned of 1 and 0 points, respectively. The total score is obtained by adding the values of the responses to the 14 items. Participants were classified into three categories of adherence to the Mediterranean diet:
* High adherence: ≥9 points
* Intermediate adherence: 7-8 points
* Low adherence: ≤6 points
* Dietary Habits Survey: This is a valid and reliable tool designed to collect information on participants' dietary practices and behaviours. It focuses on key aspects such as meal frequency, consumption of specific foods (healthy or unhealthy), cooking methods, meal times, satisfaction and desire for improvement, as well as food preferences and restrictions. The survey format was structured with closed-ended multiple-choice questions, allowing for easy analysis and comparison of responses. Clear and accessible language was used to ensure that participants understood all questions. This type of survey is useful in nutrition and public health research or intervention studies that seek to analyse the relationship between dietary habits and other factors, such as physical health, well-being or performance in older adults. High test-retest reliability (CCI > 0.80).

Laboratory analysis:

* Markers of oxidative stress.
* Markers of inflammation. Statistical analysis: statistical analysis was performed using IBM SPSS Statistics (version 28.0. Armonk, New York: IBM Corp.). Data were presented as mean ± standard deviation from the mean (SD). The level of significance was set at 95% (P=0.05). The percentage change in each variable during the different periods was calculated as Δ (%): ((post - pre) /pre × 100). Both the normality of the data and the homogeneity of the variance were checked. Once this was confirmed, a two-way ANOVA was performed to examine the time × treatment group interactions (t × g) between the two groups. As age and training are factors that influence strength and physical performance variables, they were included as possible confounding factors in the different analyses. To avoid type I errors, post hoc comparisons (pre vs. post per group) were performed. The 95% confidence interval (95% CI) and statistical power were also calculated. Differences between study periods in each experimental situation were determined using a paired sample t-test or the Wilcoxon test. Differences in Δ (%) and other tests in each study period were tested between treatment groups using the independent samples t-test or the Mann-Whitney U test with the treatment group as a fixed factor. In addition, relationships between variables were explored to perform regressions, helping us understand and predict the improvement of some variables based on others. These analyses were carried out separately for men and women to evaluate possible sex differences in the effects.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be age between 55 and 80 years.
* All individuals over the age of 55 who performed Integral Physical Conditioning training for a minimum of 120 minutes per week.
* They did not take the study supplement or any other supplement related to performance or muscle development.
* Voluntarily agreeing to participate in the study and having signed the informed consent.
* Not suffering any physical impediment to perform multicomponent physical exercise.

Exclusion Criteria:

* All individuals who were not in the age range studied.
* They did not meet the minimum weekly Comprehensive Physical Conditioning training requirement.
* All those who had suffered from or were being treated for heart, liver or kidney conditions.
* Those who were being treated with NSAIDs.
* Those who refused to stop taking supplements and/or follow the study protocol.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-11-08 (Actual); Primary Completion 2025-02-22 (Actual); Study Completion 2025-02-22 (Actual)

PRIMARY OUTCOMES:
Body composition (Day 0 and at 6 weeks of intervention). | 6 weeks
  The evaluation of body composition was performed by a dietician-nutritionist of the research group at each control point. Prior to the other tests, participants was weighed and measured by seaside telescopic staghater MOD 220. A bioelectrical impedance analysis (BIA) of body composition was also performed to minimize the effect of hydration status on all measurements. Participants was instructed to refrain from caffeine and alcohol 24 h before, as well as, if performed 12 h before the test according to published guidelines for BIA.
  To predict the MMEA, a tanita TA-MC580- 1 PLUS impedance meter (Tanita Europe B.V., UK) will be used according to the manufacturer's guidelines. The MMEA was predicted through the Equation of Sergi et al, (80): MMEA (kg) = -3.964 + (0.227 RI) + (0.095 * body mass) + (1.384 * sex) + (0.064 * XC), where RI is the standardized resistance for height and XC is the reactance.
Body composition (Day 0 after 3 weeks washout and at 6 weeks of intervention). | 6 weeks
  The evaluation of body composition was performed by a dietician-nutritionist of the research group at each control point. Prior to the other tests, participants was weighed and measured by seaside telescopic staghater MOD 220. A bioelectrical impedance analysis (BIA) of body composition was also performed to minimize the effect of hydration status on all measurements. Participants was instructed to refrain from caffeine and alcohol 24 h before, as well as, if performed 12 h before the test according to published guidelines for BIA.
  To predict the MMEA, a tanita TA-MC580- 1 PLUS impedance meter (Tanita Europe B.V., UK) will be used according to the manufacturer's guidelines. The MMEA was predicted through the Equation of Sergi et al, (80): MMEA (kg) = -3.964 + (0.227 RI) + (0.095 * body mass) + (1.384 * sex) + (0.064 * XC), where RI is the standardized resistance for height and XC is the reactance.
Nutritional evaluation (Day 0 and at 6 weeks of intervention). | 6 weeks
  The nutritional evaluation was performed by a dietitian-nutritionist of the research group at each control point. The nutritional analysis of the participants was performed using a multidimensional approach that included both food consumption frequency (T1 and T4) and adherence to the Mediterranean diet (T1, T2, T3, T4) and dietary habits (T1 and T4). The participants' dietary data were obtained through surveys and interviews, which provided information on the frequency and quantity of key food consumption. The content of macronutrients (carbohydrates, proteins and fats) and micronutrients (vitamins and minerals) was analysed, as well as the consumption patterns of foods rich in antioxidants, healthy fats and fibre.
Nutritional evaluation (Day 0 after 3 weeks washout and at 6 weeks of intervention). | 6 weeks
  The nutritional evaluation was performed by a dietitian-nutritionist of the research group at each control point. The nutritional analysis of the participants was performed using a multidimensional approach that included both food consumption frequency (T1 and T4) and adherence to the Mediterranean diet (T1, T2, T3, T4) and dietary habits (T1 and T4). The participants' dietary data were obtained through surveys and interviews, which provided information on the frequency and quantity of key food consumption. The content of macronutrients (carbohydrates, proteins and fats) and micronutrients (vitamins and minerals) was analysed, as well as the consumption patterns of foods rich in antioxidants, healthy fats and fibre.
Assessment of muscle strength and performance. Short Physical Performance Battery (Day 0 and at 6 weeks of intervention). | 6 weeks
  Short Physical Performance Battery (SPPB): consists of 3 tests to be used to assess lower extremity function following standard protocols:
  * Balance by balance test.
  * Muscle strength test in the legs, sit to up test.
  * Mobility test using gait speed, gait speed test. It is important to follow the sequence of the tests, because if the patient starts to stand and sit, he/she may become fatigued and perform falsely poorly in the other two tests. The average test duration is between 6 and 10 min. Each test will be scored from 0 to 4. A score of 0 represent an inability to complete the test, and a score of 4 represent the highest level of performance. Therefore, total scores (SPPB scores) range from 0 to 12, and a higher SPPB score indicate a higher level of physical fitness.
Assessment of muscle strength and performance. Short Physical Performance Battery (Day 0 after 3 weeks washout and at 6 weeks of intervention). | 6 weeks
  Short Physical Performance Battery (SPPB): consists of 3 tests to be used to assess lower extremity function following standard protocols:
  * Balance by balance test.
  * Muscle strength test in the legs, sit to up test.
  * Mobility test using gait speed, gait speed test. It is important to follow the sequence of the tests, because if the patient starts to stand and sit, he/she may become fatigued and perform falsely poorly in the other two tests. The average test duration is between 6 and 10 min. Each test will be scored from 0 to 4. A score of 0 represent an inability to complete the test, and a score of 4 represent the highest level of performance. Therefore, total scores (SPPB scores) range from 0 to 12, and a higher SPPB score indicate a higher level of physical fitness.
Assessment of muscle strength and performance. Timed-up-and-go (Day 0 and at 6 weeks of intervention). | 6 weeks
  The evaluation of muscular strength and physical performance was performed by a strength and conditioning coach graduated in physical activity and sport sciences, which was carried out at each control point. The tests to be performed to the participants was:
  Timed-up-and-go (TUG): Timed-up-and-go is used to assess mobility, balance and agility. Participants are instructed to get up from a chair without assistance (starting point), walk forward three meters (m), walk back to the chair and sit down again (end of test). They are asked to perform the test at a normal, everyday pace, using marks on the floor to indicate where to turn. The total time used from the beginning to the end of the test is recorded.
Assessment of muscle strength and performance. Timed-up-and-go (Day 0 after 3 weeks washout and at 6 weeks of intervention). | 6 weeks
  The evaluation of muscular strength and physical performance was performed by a strength and conditioning coach graduated in physical activity and sport sciences, which was carried out at each control point. The tests to be performed to the participants was:
  Timed-up-and-go (TUG): Timed-up-and-go is used to assess mobility, balance and agility. Participants are instructed to get up from a chair without assistance (starting point), walk forward three meters (m), walk back to the chair and sit down again (end of test). They are asked to perform the test at a normal, everyday pace, using marks on the floor to indicate where to turn. The total time used from the beginning to the end of the test is recorded.
Assessment of muscle strength and performance. 400-meter Walk Test Perfomance (Day 0 and at 6 weeks of intervention). | 6 weeks
  The evaluation of muscular strength and physical performance was performed by a strength and conditioning coach graduated in physical activity and sport sciences, which will be carried out at each control point. The tests to be performed to the participants was:
  400-meter Walk Test Perfomance: measures mobility and cardiovascular fitness through a 400-meter timed walk (min). Cones are placed 20 m apart, around which participants must move 10 times, back and forth, as fast as possible. Only one attempt was allowed.
Assessment of muscle strength and performance. 400-meter Walk Test Perfomance (Day 0 after 3 weeks washout and at 6 weeks of intervention). | 6 weeks
  The evaluation of muscular strength and physical performance was performed by a strength and conditioning coach graduated in physical activity and sport sciences, which will be carried out at each control point. The tests to be performed to the participants was:
  400-meter Walk Test Perfomance: measures mobility and cardiovascular fitness through a 400-meter timed walk (min). Cones are placed 20 m apart, around which participants must move 10 times, back and forth, as fast as possible. Only one attempt was allowed.
Assessment of muscle strength and performance. Grip strength (Day 0 and at 6 weeks of intervention). | 6 weeks
  The evaluation of muscular strength and physical performance was performed by a strength and conditioning coach graduated in physical activity and sport sciences, which will be carried out at each control point. The tests to be performed to the participants was:
  Grip strength: isometric hand strength is a commonly used measure to establish upper body skeletal muscle function and has been widely used as a general indicator of physical fitness. Grip strength was measured using a validated hydraulic hand-held dynamometer (Jamar plus +, if instruments, Adelaide, Australia). Values will be recorded in kilograms. Grip strength will be measured while seated, elbow in 90° flexion and wrist in neutral position. Participants was asked to apply maximum grip strength in 3 different attempts with the left and right hands. Between each attempt, a 30 s rest was allowed. The measurement in which the maximum grip strength is obtained from the 3 attempts will be used.
Assessment of muscle strength and performance. Grip strength (Day 0 after 3 weeks washout and at 6 weeks of intervention). | 6 weeks
  The evaluation of muscular strength and physical performance was performed by a strength and conditioning coach graduated in physical activity and sport sciences, which will be carried out at each control point. The tests to be performed to the participants was:
  Grip strength: isometric hand strength is a commonly used measure to establish upper body skeletal muscle function and has been widely used as a general indicator of physical fitness. Grip strength was measured using a validated hydraulic hand-held dynamometer (Jamar plus +, if instruments, Adelaide, Australia). Values will be recorded in kilograms. Grip strength will be measured while seated, elbow in 90° flexion and wrist in neutral position. Participants was asked to apply maximum grip strength in 3 different attempts with the left and right hands. Between each attempt, a 30 s rest was allowed. The measurement in which the maximum grip strength is obtained from the 3 attempts will be used.
Isometric strength of legs and back (Day 0 and at 6 weeks of intervention) | 6 Weeks
  A BASELINE traction dynamometer (back and leg dynamometer) with adjustable handle and base platform was used. The objective was to assess the maximum isometric strength of the back and leg extensor muscles (kg).
  The subject stood with their feet shoulder-width apart on the dynamometer platform. The legs were slightly bent and the back was in a neutral, inclined position. The dynamometer was adjusted so that the subject could grasp the handle with their arms fully extended downwards (near the knees). The subject was asked to pull the handle upwards, using their back and leg strength, without bending their arms or leaning their trunk backwards. The movement was isometric; force was applied without visible displacement. The contraction lasted about 3 to 5 seconds. Two attempts were made with at least 30 seconds of rest between them. The maximum value achieved was recorded.
Isometric strength of legs and back (Day 0 after 3 weeks washout and at 6 weeks of intervention). | 6 Weeks
  A BASELINE traction dynamometer (back and leg dynamometer) with adjustable handle and base platform was used. The objective was to assess the maximum isometric strength of the back and leg extensor muscles (kg).
  The subject stood with their feet shoulder-width apart on the dynamometer platform. The legs were slightly bent and the back was in a neutral, inclined position. The dynamometer was adjusted so that the subject could grasp the handle with their arms fully extended downwards (near the knees). The subject was asked to pull the handle upwards, using their back and leg strength, without bending their arms or leaning their trunk backwards. The movement was isometric; force was applied without visible displacement. The contraction lasted about 3 to 5 seconds. Two attempts were made with at least 30 seconds of rest between them. The maximum value achieved was recorded.
Isometric arm flexion strength (Day 0 and at 6 weeks of intervention) | 6 Weeks
  A BASELINE traction dynamometer with adjustable handle and base platform was used. The objective was to assess the maximum isometric strength of the upper body (kg), specifically the arm flexor muscles (biceps). The subject stood with their feet shoulder-width apart on the dynamometer platform. Their legs were slightly bent and their back was straight and upright. The dynamometer was adjusted so that the subject could grasp the handle with their arms bent at 90°, elbows close to the body and wrists in a supine position. The subject was asked to pull the handle upwards, exerting force with their arms, without leaning the trunk backwards or using momentum. The movement was isometric; force was applied without visible displacement. The contraction lasted about 3 to 5 seconds. Two attempts were made with a 30-second rest between them. The maximum value achieved was recorded
Isometric arm flexion strength (Day 0 after 3 weeks washout and at 6 weeks of intervention) | 6 Weeks
  A BASELINE traction dynamometer with adjustable handle and base platform was used. The objective was to assess the maximum isometric strength of the upper body (kg), specifically the arm flexor muscles (biceps). The subject stood with their feet shoulder-width apart on the dynamometer platform. Their legs were slightly bent and their back was straight and upright. The dynamometer was adjusted so that the subject could grasp the handle with their arms bent at 90°, elbows close to the body and wrists in a supine position. The subject was asked to pull the handle upwards, exerting force with their arms, without leaning the trunk backwards or using momentum. The movement was isometric; force was applied without visible displacement. The contraction lasted about 3 to 5 seconds. Two attempts were made with a 30-second rest between them. The maximum value achieved was recorded
30-second push-up test (Day 0 and at 6 weeks of intervention) | 6 Weeks
  This test was performed to assess the muscle strength and endurance (push) of the upper body (mainly pectorals, deltoids and triceps) and the stabilising strength of the lumbar-abdominal girdle. It consisted of performing as many push-ups as possible in 30 seconds from a plank position. The participant is placed in a high plank position with arms extended, hands shoulder-width apart, and body aligned from ankles to head. Each push-up must be performed with a full range of motion: lower the chest close to the floor (about 5-8 cm) and fully extend the elbows when rising. Only correctly executed repetitions were counted and recorded.
30-second push-up test (Day 0 after 3 weeks washout and at 6 weeks of intervention) | 6 Weeks
  This test was performed to assess the muscle strength and endurance (push) of the upper body (mainly pectorals, deltoids and triceps) and the stabilising strength of the lumbar-abdominal girdle. It consisted of performing as many push-ups as possible in 30 seconds from a plank position. The participant is placed in a high plank position with arms extended, hands shoulder-width apart, and body aligned from ankles to head. Each push-up must be performed with a full range of motion: lower the chest close to the floor (about 5-8 cm) and fully extend the elbows when rising. Only correctly executed repetitions were counted and recorded.
30-second supine trunk flexion test (Day 0 and at 6 weeks of intervention) | 6 Weeks
  Crunch Test: the objective was to assess abdominal muscle endurance. The subject lay supine with knees bent at 90° and feet flat on the floor and arms crossed over the chest. At the evaluator's signal, the subject performed as many trunk flexions as possible in 30 seconds. A repetition was counted as valid when the shoulders clearly lifted off the floor without lifting the lower back and returned to the starting position. The total number of correct repetitions was recorded.
30-second supine trunk flexion test (0 day after 3 weeks washout and at 6 weeks of intervention) | 6 Weeks
  Crunch Test: the objective was to assess abdominal muscle endurance. The subject lay supine with knees bent at 90° and feet flat on the floor and arms crossed over the chest. At the evaluator's signal, the subject performed as many trunk flexions as possible in 30 seconds. A repetition was counted as valid when the shoulders clearly lifted off the floor without lifting the lower back and returned to the starting position. The total number of correct repetitions was recorded.
Isometric pull-up strength test (Day 0 and at 6 weeks of intervention) | 6 Weeks
  Flexed Arm Hang Test: used to assess the isometric strength and muscular endurance of the upper body, especially the arms, shoulders and back. Hanging from the bar, keep your head above the bar for as long as possible. The subject stands under a fixed horizontal bar, such as a pull-up bar. With the help of a bench or assistance, they position themselves with their elbows bent and their chin above the level of the bar. The palms may be pronated. The stopwatch starts when the person is suspended without assistance, with their feet completely off the ground. The test ends when the chin falls below the bar, the arms are extended, or the subject lets go.
Isometric pull-up strength test (Day 0 after 3 weeks washout and at 6 weeks of intervention) | 6 Weeks
  Flexed Arm Hang Test: used to assess the isometric strength and muscular endurance of the upper body, especially the arms, shoulders and back. Hanging from the bar, keep your head above the bar for as long as possible. The subject stands under a fixed horizontal bar, such as a pull-up bar. With the help of a bench or assistance, they position themselves with their elbows bent and their chin above the level of the bar. The palms may be pronated. The stopwatch starts when the person is suspended without assistance, with their feet completely off the ground. The test ends when the chin falls below the bar, the arms are extended, or the subject lets go.
Seated dumbbell arm curl test (Day 0 and at 6 weeks of intervention) | 6 Weeks
  The dynamic strength of the arm flexor muscles was measured. The participant sat on a chair without armrests, with their back straight and their feet flat on the floor. They held a dumbbell in their dominant hand with their palm facing upwards and their arm fully extended down at their side. In 30 seconds, the participant completely flexed their elbow, bringing the dumbbell towards their chest without moving their shoulder, and then extended it again.
  Complete repetitions were counted. A 2 kg dumbbell was used for women and a 4 kg dumbbell for men.
Seated dumbbell arm curl test (Day 0 after 3 weeks washout and at 6 weeks of intervention) | 6 Weeks
  The dynamic strength of the arm flexor muscles was measured. The participant sat on a chair without armrests, with their back straight and their feet flat on the floor. They held a dumbbell in their dominant hand with their palm facing upwards and their arm fully extended down at their side. In 30 seconds, the participant completely flexed their elbow, bringing the dumbbell towards their chest without moving their shoulder, and then extended it again.
  Complete repetitions were counted. A 2 kg dumbbell was used for women and a 4 kg dumbbell for men.
Quality of Life Assessment (Day 0 and at 6 weeks of intervention) | 6 weeks
  The WHOQOL-BREF test was used in all controls. This questionnaire is a shortened version of the WHOQOL-100 questionnaire, developed by the World Health Organisation (WHO) to assess quality of life. It is one of the most widely used instruments internationally due to its psychometric robustness, cross-cultural applicability and brevity.There were 26 questions divided into 4 domains (Physical, Phychological, Social and Enviromental). Plus 2 questions on perception of quality of life and health that were not counted.
Quality of Life Assessment (Day 0 after 3 weeks washout and at 6 weeks of intervention) | 6 weeks
  The WHOQOL-BREF test was used in all controls. This questionnaire is a shortened version of the WHOQOL-100 questionnaire, developed by the World Health Organisation (WHO) to assess quality of life. It is one of the most widely used instruments internationally due to its psychometric robustness, cross-cultural applicability and brevity.There were 26 questions divided into 4 domains (Physical, Phychological, Social and Enviromental). Plus 2 questions on perception of quality of life and health that were not counted.
Inflammation markers. CRP (Day 0 and at 6 weeks of intervention). | 6 weeks
  CRP was assessed in duplicate from frozen stored serum. PCR levels using an enzyme-linked immunostorbent assay based on purified proteins and purified anti-CRP antibodies (Calbiochem, San Diego, CA).
Inflammation markers. CRP(Day 0 after 3 weeks washout and at 6 weeks of intervention). | 6 weeks
  CRP was assessed in duplicate from frozen stored serum. PCR levels using an enzyme-linked immunostorbent assay based on purified proteins and purified anti-CRP antibodies (Calbiochem, San Diego, CA).
Inflammation markers. Cytokine levels and cytokine soluble receptors (Day 0 and at 6 weeks of intervention). | 6 weeks
  IL-1 (soluble IL-1 receptor [IL-1SR]), IL-2 (soluble IL-2 receptor [il-2SR]), IL-6 (soluble IL-6 receptor [IL-6SR]), IL-7 (soluble IL-7 receptor [IL-7SR]) was measured using enzyme-linked immunostorbent assay kits (Research and Development Systems, Minneapolis, MN).
Inflammation markers. Cytokine levels and cytokine soluble receptors (Day 0 after 3 weeks washout and at 6 weeks of intervention). | 6 weeks
  IL-1 (soluble IL-1 receptor [IL-1SR]), IL-2 (soluble IL-2 receptor [il-2SR]), IL-6 (soluble IL-6 receptor [IL-6SR]), IL-7 (soluble IL-7 receptor [IL-7SR]) was measured using enzyme-linked immunostorbent assay kits (Research and Development Systems, Minneapolis, MN).
Inflammation markers. TNF-α (Day 0 and at 6 weeks of intervention). | 6 weeks
  TNF-α (TNFSR1 and TNFSR2) levels was assessed in duplicate from frozen stored serum.
Inflammation markers. TNF-α (Day 0 after 3 weeks washout and at 6 weeks of intervention). | 6 weeks
  TNF-α (TNFSR1 and TNFSR2) levels was assessed in duplicate from frozen stored serum.
Oxidative stress markers. Reduced (GSH) and oxidized glutathione (GSSG) (Day 0 and at 6 weeks of intervention). | 6 weeks
  Reduced (GSH) and oxidized glutathione (GSSG) was determined using colorimetric kits. Reducing power will be calculated by the equation GSH/(GSH + GSSG).
Oxidative stress markers. Reduced (GSH) and oxidized glutathione (GSSG) (Day 0 after 3 weeks washout and at 6 weeks of intervention). | 6 weeks
  Reduced (GSH) and oxidized glutathione (GSSG) was determined using colorimetric kits. Reducing power will be calculated by the equation GSH/(GSH + GSSG).
Oxidative stress markers. TBAR (Day 0 and at 6 weeks of intervention). | 6 weeks
  Lipid peroxidation was analyzed in plasma as thiobarbituric acid reactive substances (TBAR). The TBAR was determined after treatment of the sample with 4% butylated hydroxytoluene and an additional reaction with 0.375% thiobarbituric acid in 0.25 M HCl and 1% Triton X-100 (15 min, at 100°C).
Oxidative stress markers. TBAR (Day 0 after 3 weeks washout and at 6 weeks of intervention). | 6 weeks
  Lipid peroxidation was analyzed in plasma as thiobarbituric acid reactive substances (TBAR). The TBAR was determined after treatment of the sample with 4% butylated hydroxytoluene and an additional reaction with 0.375% thiobarbituric acid in 0.25 M HCl and 1% Triton X-100 (15 min, at 100°C).
Oxidative stress markers. Malondialdehye equivalents (MDA) (Day 0 and at 6 weeks of intervention). | 6 weeks
  Malondialdehye equivalents (MDA) was calculated according to the absorbance at 535 nm against a blank (lacking TBA) and using 1,1,2,2-tetroxyethylpropane as standard.
Oxidative stress markers. Malondialdehye equivalents (MDA) (Day 0 after 3 weeks washout and at 6 weeks of intervention). | 6 weeks
  Malondialdehye equivalents (MDA) was calculated according to the absorbance at 535 nm against a blank (lacking TBA) and using 1,1,2,2-tetroxyethylpropane as standard.
Oxidative stress markers. Superoxide dismutase (SOD) (Day 0 and at 6 weeks of intervention). | 6 weeks
  Superoxide dismutase (SOD) was estimated by inhibition of adrenaline autooxidation, read at 480 nm in a spectrophotometer.
Oxidative stress markers. Superoxide dismutase (SOD) (Day 0 after 3 weeks washout and at 6 weeks of intervention). | 6 weeks
  Superoxide dismutase (SOD) was estimated by inhibition of adrenaline autooxidation, read at 480 nm in a spectrophotometer.
Oxidative stress markers. Nitric oxide (NO) (Day 0 and at 6 weeks of intervention). | 6 weeks
  Nitric oxide (NO) was estimated spectrophotometrically as a function of nitrite generation.
Oxidative stress markers. Nitric oxide (NO) (Day 0 after 3 weeks washout and at 6 weeks of intervention). | 12 weeks
  Nitric oxide (NO) was estimated spectrophotometrically as a function of nitrite generation.
Oxidative stress markers. Total antioxidant capacity (TAC) (Day 0 and at 6 weeks of intervention). | 6 weeks
  Total antioxidant capacity (TAC) was analyzed in duplicate samples, and absorbance will be measured using a microplate reader.
Oxidative stress markers. Total antioxidant capacity (TAC) (Day 0 after 3 weeks washout and at 6 weeks of intervention). | 6 weeks
  Total antioxidant capacity (TAC) was analyzed in duplicate samples, and absorbance will be measured using a microplate reader.
Hormones. Total serum testosterone (Day 0 and at 6 weeks of intervention). | 6 weeks
  Total serum testosterone was measured using the enzyme from commercially available enzyme-linked immunosorbent assay (ELISA) kits (DRG Testosterone ELISA KIT, DRG Instruments GmbH, Marburg,® Germany).
Hormones. Total serum testosterone (Day 0 after 3 weeks washout and at 6 weeks of intervention).. | 6 weeks
  Total serum testosterone was measured using the enzyme from commercially available enzyme-linked immunosorbent assay (ELISA) kits (DRG Testosterone ELISA KIT, DRG Instruments GmbH, Marburg,® Germany).
Hormones. Sex hormone binding globulin (SHBG) (Day 0 and at 6 weeks of intervention). | 6 weeks
  Sex hormone binding globulin (SHBG) was measured by chemiluminescence based on the immunometric method (immunite, 2000), which will be from the same supplier as testosterone.
Hormones. Sex hormone binding globulin (SHBG) (Day 0 after 3 weeks washout and at 6 weeks of intervention). | 6 weeks
  Sex hormone binding globulin (SHBG) was measured by chemiluminescence based on the immunometric method (immunite, 2000), which will be from the same supplier as testosterone.
Hormones. Cortisol (Day 0 and at 6 weeks of intervention). | 6 weeks
  Cortisol was measured by enzyme-linked fluorescent assay in a microplate reader (Cytation 5 Cell Imaging Multi-Mode Reader -Biotek Instruments, USA).
Hormones. Cortisol (Day 0 after 3 weeks washout and at 6 weeks of intervention). | 6 weeks
  Cortisol was measured by enzyme-linked fluorescent assay in a microplate reader (Cytation 5 Cell Imaging Multi-Mode Reader -Biotek Instruments, USA).
Hormones. Total testosterone/cortisol and total testosterone/SHBG ratios (Day 0 and at 6 weeks of intervention). | 6 weeks
  Total testosterone/cortisol and total testosterone/SHBG ratios was calculated from serum testosterone, cortisol and SHBG concentrations.
Hormones. Total testosterone/cortisol and total testosterone/SHBG ratios (Day 0 after 3 weeks washout and at 6 weeks of intervention). | 6 weeks
  Total testosterone/cortisol and total testosterone/SHBG ratios was calculated from serum testosterone, cortisol and SHBG concentrations.

CONTACTS AND LOCATIONS:
Locations (1):
- Juan Mielgo Ayuso, Burgos, Burgos, Spain

IPD SHARING:
Plan to Share IPD: No